CLINICAL TRIAL: NCT03064542
Title: The Role of Thyroid Status in Regulating Brown Adipose Tissue Activity, White Adipose Tissue Partitioning and Resting Energy Expenditure
Acronym: TRIBUTE
Status: Completed | Type: Observational
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Agency for Science, Technology and Research (Other)
Responsible Party: Principal Investigator, Melvin Leow, Principal Investigator, Tan Tock Seng Hospital
Other Study IDs: 2015/00718
Record Dates: First submitted 2017-02-09; First posted 2017-02-27 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism | interventions — Carbimazole; Methimazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood samples for thyroid function, liver and kidney function, fasting glucose, insulin and lipids, analysis of fat metabolism and protein profiles.
  Urine samples for fat metabolism and protein profiles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: carbimazole (CMZ) or thiamazole (TMZ) — CMZ or TMZ will be used to treat the hyperthyroidism till the FT4/TSH is in normal range.

SUMMARY:
To determine how thyroid status regulates the relationship between brown adipose tissue (BAT) volume/activity, white adipose tissue (WAT) partitioning and basal metabolic rate (BMR) in hyperthyroid patients transitioning to euthyroidism via antithyroid drugs.

To compare euthyroid outcomes (BAT, WAT, BMR, body composition, body weight and insulin resistance) achieved by hypothalamus-pituitary-thyroid (HPT) set point vs. normal ranges of plasma free thyroxine 4 (FT4) and throxine stimulating hormone (TSH).

DETAILED DESCRIPTION:
Study Visit 1 is meant to confirm if subject's hyperthyroidism is due to Graves' disease via a blood test called TSH receptor autoantibody (TRAb). This is a standard test that the doctor will routinely order as part of clinical practice to diagnose the cause of the subject's hyperthyroidism and is not part of the research procedure. If this TRAb blood test has been done before the subjects have been referred to the endocrinology clinic at TTSH, the doctors will review that result and decide if a repeat test is needed. If subjects are confirmed by blood tests to have Graves' disease type of hyperthyroidism, they are eligible to take part in this study. However, approximately 2 teaspoons (~ 10 mL) of blood will be taken for baseline thyroid function test just prior to the initiation of anti-thyroid drugs. Pre-menopausal women will also undergo a urine pregnancy test to exclude pregnancy prior to participation at study entry. Once subjects have consented to participate in this study, they will receive standard antithyroid drug (ATD) therapy as indicated clinically which in current practice will either be carbimazole (CMZ) or thiamazole (TMZ).The clinic endocrinologists at TTSH will be in charge of deciding on the ATD dose required based on the latest FT4, FT3 and TSH blood test results as per standard medical practice. . Subjects will then be scheduled for Visit 2 for baseline research measurements while you are still hyperthyroid.

On Study Visit 2, subjects will be asked to come to the Clinical Nutrition Research Centre (CNRC) at the Centre for Translational Medicine at the National University of Singapore in the morning at 0830 h after an overnight fast of 8-10 hours. Subjects will undergo anthropometry (ie. measures of body weight, height, waist and hip circumference), non-invasive percentage fat estimation using bioelectrical impedence analysis (BIA) and body composition evaluation using dual energy X-ray absorptiometry (DXA) which allows quantification of fat, lean and bone mass. Subjects will then undergo metabolic rate measurement in a whole body calorimeter coupled with infrared thermography using a thermal camera mounted on a tripod stand (IRT) focusing on the neck and area above the collar bone in a whole body room calorimeter for the next 45 minutes.

Subjects will then proceed to the Clinical Imaging Research Centre (CIRC) also located in the same building at the basement where an intravenous indwelling cannula will be inserted into an arm vein from which a fasting blood sample will be taken. At first, 30 mL of blood will be taken (about 6 teaspoons) in which 10 mL will be tested for thyroid function while the other 10 mL will be tested for liver and kidney function and the remaining 10mL for fasting glucose, insulin and lipids. An additional 20 mL blood (about 4 teaspoons) will be taken for analysis of markers of fat metabolism and protein profiles reflective of brown fat activity. A urine sample will also be collected. Subsequently, subjects will be given an intravenous injection of a radioactive labeled glucose called 18-FDG through the intravenous cannula and followed by PET and fat fraction MRI scanning for BAT and MRI-MRS of abdominal white fat for the next 1 hour.

After that, subjects will then be required to go to the endocrinology clinic at TTSH for control of their hyperthyroidism via ATD. This may take about 6 months to attain stable thyroid hormones levels (FT4, FT3, TSH). Subjects will be followed up every 6-8 weeks as per standard medical practice by theTTSH endocrinologist and have their ATD doses adjusted till their thyroid function tests are stable'. When this happens, subjects will continue with the remaining part of the research, which is Study Visit 3. With the exception an additional urine pregnancy test, Study Visit 3 is exactly the same as Study Visit 2.

ELIGIBILITY:
Inclusion Criteria:

* You must be aged 21 to 50 years old (no gender restrictions).
* You must be diagnosed with Graves' disease.
* You are able to give informed consent..
* You must have body mass index (BMI) between 18.5 to 29.9 kg/m2 inclusive.
* You must be treated with carbimazole (CMZ) or thiamazole (TMZ) and compliant to treatment.
* Willing to avail yourself for the whole study and follow study procedures.

Exclusion Criteria:

* Chronic illnesses such as diabetes mellitus or cancer.
* You have a known history of liver or kidney disease.
* Female subjects who are pregnant or contemplating pregnancy.
* Those allergic to carbimazole (CMZ) or thiamazole (TMZ).
* History of surgery with metallic clips, staples or stents.
* Those on drugs that might affect body composition (eg. steroids) or BAT (eg. beta-blockers).
* Those with poor compliance to medication.
* Presence of cardiac pacemaker or other foreign body in any part of the body.
* History of claustrophobia particularly in a MRI scanner.
* Those with a history of bronchial asthma.
* Those with overt congestive heart failure.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Hyperthyroid patients diagnosed with Graves' disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Thyroid function test (serum free thyroxine (FT4) and serum thyroid stimulating hormone (TSH). | 6 months of treatment with an anti-thyroid drug
  This observation supports the concept of a unique set point in FT4 and TSH for any given individual and forms the basis for optimization of thyroid status by targeting the FT4 and TSH levels towards the set point. All data, study and clinical endpoints will be analyzed and correlated by the proximity of the final stable euthyroid Thyroid function test (TFT) to the predicted euthyroid set point using the computer software.

SECONDARY OUTCOMES:
Fat volume- Brown adipose tissue (BAT) | 6 months of treatment with an anti-thyroid drug
  The above volumes will be measured at start of treatment and at 6 months by MRI (fat fraction for BAT) - volumes in mL.
Fat volume- White adipose tissue (WAT) | 6 months of treatment with an anti-thyroid drug
  The above volumes will be measured at start of treatment and at 6 months by MRI (standard MRI for WAT) - volumes in mL.
Energy expenditure | 6 months of treatment with an anti-thyroid drug
  The metabolic rate (measured from the energy expenditure) will be measured using the whole body calorimeter in kcal/day.
Body composition | 6 months of treatment with an anti-thyroid drug
  The subjects will have a body composition evaluated by DXA at the start of treatment and 6 months post-treatment when they are rendered euthyroid. WE will measure lean mass, fat mass and bone mass.
Infrared thermography (IRT) | 6 months of treatment with an anti-thyroid drug
  We will measure BAT activity using IRT. This will be expressed in terms of temperature change in degrees Celsius and heat power change in watts (W).

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Endocrinology Clinic, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun L, Goh HJ, Verma S, Govindharajulu P, Sadananthan SA, Michael N, Henry CJ, Goh JP, Velan SS, Leow MK. Brown adipose tissues mediate the metabolism of branched chain amino acids during the transitioning from hyperthyroidism to euthyroidism (TRIBUTE). Sci Rep. 2022 Mar 7;12(1):3693. doi: 10.1038/s41598-022-07701-7. PMID 35256693